CLINICAL TRIAL: NCT03100877
Title: Phase I-II Single Cycle Melphalan/Total Marrow Irradiation (TMI) and Autologous Stem Cell Transplantation (ASCT) Followed by Maintenance in Patients With High-Risk Myeloma and/or Poor Response to Induction Therapy Within 12 Months of Diagnosis
Brief Title: Melphalan, Total Marrow Irradiation, and Autologous Stem Cell Transplantation in Treating Patients With High-Risk Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Feasibility Issues
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16464; NCI-2017-00512 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16464 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Plasma Cell Leukemia in Remission; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Lenalidomide; Blood Component Removal; Leukapheresis; Melphalan; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mel/TMI, ASCT) (Experimental): MOBILIZATION AND APHERESIS: Patients receive cyclophosphamide IV over 2 hours. Beginning 24 hours after cyclophosphamide administration, patients receive filgrastim SC or IV. Patients also undergo apheresis over 4 hours on day 10.
  CONDITIONING REGIMEN: Patients receive palifermin IV on days -8, to -6, undergo TMI on days -5 to -2, and receive melphalan IV over 30 minutes on day -1. Patients then undergo ASCT IV on day 0, receive palifermin IV on days 1-3, and receive filgrastim SC or IV on day 5.
  MAINTENANCE THERAPY: Beginning 30 days after ASCT, patients receive lenalidomide PO daily.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Procedure: pheresis; Drug: Melphalan; Biological: Palifermin; Radiation: Total Marrow Irradiation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Autologous Stem Cell Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: pheresis — Undergo apheresis
  Other Names: leukapheresis; Leukocytopheresis; Therapeutic Leukopheresis; apheresis
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Palifermin — Given IV
  Other Names: Growth Factor, Recombinant Human Keratinocyte; Kepivance; Keratinocyte Growth Factor, Recombinant Human; Recombinant Human Keratinocyte Growth Factor; rhKGF; rhu Keratinocyte Growth Factor
Radiation: Total Marrow Irradiation — Undergo TMI

SUMMARY:
This phase I/II trial studies the side effects and best dose of melphalan and total marrow irradiation and how well they work with autologous stem cell transplantation in treating patients with high-risk multiple myeloma. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Total marrow irradiation is a type of radiation therapy and a form of total body irradiation that may deliver focused radiation to the major marrow sites where cancer cells reside. Giving chemotherapy and total-body irradiation before a peripheral autologous blood stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and determine the maximum tolerated dose (MTD) of melphalan and fractionated total marrow irradiation (TMI) as conditioning regimen for autologous stem cell transplantation (ASCT) in patients with high-risk or treatment-insensitive multiple myeloma (MM). (Phase I) II. Evaluate the safety of the regimen at each dose level by assessing adverse events: type, frequency, severity, attribution, time course, duration.

III. Evaluate the safety of the regimen at each dose level by assessing complication including: infection, delayed engraftment and secondary malignancy.

IV. To assess complete response (CR) and minimal residual disease (MRD) rates at 100 days post ASCT in a phase II expanded cohort of patients treated at the MTD. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the predictive value of high risk features inclusive of fluorescent in situ hybridization (FISH), lactate dehydrogenase (LDH), International Staging System (ISS) stage, gene expression profiling (GEP) for CR and minimal residual disease (MRD) for relapse free survival/progression free survival/overall survival (RFS/PFS/OS) after melphalan TMI (mel/TMI).

II. To assess MRD by positron emission tomography (PET), next generation sequencing (NGS), and flow cytometry after mel/TMI, prior to maintenance and correlation with PFS and OS.

III. To assess in a descriptive fashion PFS and OS following mel/TMI and ASCT. IV. Evaluate changes in fludeoxyglucose F-18 (FDG) PET pre and post TMI/melphalan.

TERTIARY OBJECTIVES:

I. Assessment of bone marrow residual damage. II. Assessment of immune recovery dynamics. III. To conduct genetic profiling of myeloma cells. IV. Multimodal imaging for non-invasive assessment of treatment effect on bone and marrow.

OUTLINE: This is a phase I, dose-escalation study of melphalan and TMI followed by a phase II study.

MOBILIZATION AND APHERESIS: Patients receive cyclophosphamide intravenously (IV) over 2 hours. Beginning 24 hours after cyclophosphamide administration, patients receive filgrastim subcutaneously (SC) or IV. Patients also undergo apheresis over 4 hours on day 10.

CONDITIONING REGIMEN: Patients receive palifermin IV on days -8, to -6, undergo TMI on days -5 to -2, and receive melphalan IV over 30 minutes on day -1. Patients then undergo ASCT IV on day 0, receive palifermin IV on days 1-3, and receive filgrastim SC or IV on day 5.

MAINTENANCE THERAPY: Beginning 30 days after ASCT, patients receive lenalidomide orally (PO) daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients with will be eligible if they are either in partial response, or have stable disease after no more than two attempts of induction therapy
* Patients with high-risk cytogenetics, t(4:14); t(14;16), t(14:20), deletion p17, gain in 1q, are eligible
* Patients with plasma cell leukemia in >= partial remission are eligible
* Patients with non-quantifiable monoclonal proteins are eligible provided they meet other criteria for multiple myeloma and they have evaluable or measurable disease by other (radiographic, magnetic resonance imaging [MRI], computed tomography [CT], lytic measurable lesion on x-ray,) means
* Karnofsky performance status (KPS) >= 70%
* Less than 12 months since diagnosis
* No contraindication to the collection of a minimum of 4 x 10^6 CD34+ cells/kg by apheresis
* Bilirubin =< 1.5 mg/dl
* Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x upper limits of normal
* Creatinine of measured or calculated creatinine clearance of >= 50 cc/min
* Absolute neutrophil count of > 1000/ul
* Platelet count of > 100,000/ul
* Cardiac ejection fraction >= 50% by multi-gated acquisition (MUGA) scan and/or by echocardiogram
* Forced expiratory volume in 1 second (FEV1) > 60% and diffusion capacity of the lung for carbon monoxide (DLCO) > 50% of predicted lower limit
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately; patients must be fully aware of the teratogenic potential of immunomodulatory drugs (ImIDs) and agree to fully comply with the mandated guidelines regarding contraception as stated in the informed consent and the patient warning document attached to the consent form; women of childbearing potential must have a negative pregnancy test performed within 24 hours prior to beginning thalidomide, except for woman who have been postmenopausal for at least 2 years, or underwent hysterectomy; use of effective means of contraceptive should be started at least 2 weeks prior to initiating lenalidomide
* All subjects must have the ability to understand and the willingness to sign a written informed consent; they are to give voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Patients should have finished their prior systemic therapy or radiation therapy, at least 3 weeks before cyclophosphamide or granulocyte colony-stimulating factor (G-CSF)/plerixafor mobilization, and should have finished dexamethasone at least 7 days prior to Plerixafor priming; administration of bisphosphonates needs to be completed at least 2 weeks before cyclophosphamide priming; bisphosphonates can be resumed or started after day 30

Exclusion Criteria:

* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low-risk prostate cancer after curative therapy
* Known hypersensitivity to filgrastim or to Escherichia coli (E. coli) derived proteins
* Inability to lie supine in a full body cast for approximately 30 minutes, the anticipated duration of each treatment session
* Previous radiation therapy to more than 20% of bone marrow containing areas, or to any area exceeding 2000 cGy, is an exclusion
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* No other medical, or psychosocial problems, which in the opinion of the primary physician or principal investigator would place the patient at unacceptably high risk from this treatment regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-05-24 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) post-Autologous Stem Cell Transplantation (ASCT) (Phase II) | Up to 3 years
  Will be summarized both by pooling across dose levels and by dose level.
Maximum Tolerated Dose (MTD) of mel/TMI (Phase I) | Up to 3 years
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States